CLINICAL TRIAL: NCT00961662
Title: Dose Ranging Effects of Three Low-doses of Naturlose™ (Tagatose) on Glycemic Control and Safety of Naturlose™ (Tagatose) Over Six Months in Subjects With Mild Type 2 Diabetes Mellitus Under Control With Diet and Exercise.
Brief Title: A Clinical Study to Evaluate the Effect of Naturlose (Tagatose)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Lodder (Industry)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Robert Lodder, PhD, Spherix Incorporated
Organization: Spherix Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70971-005
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tagatose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2.5 active (Experimental): 2.5 Active - 2.5 g D-tagatose given orally, three times daily, immediately prior to meals for 6 months.
  Interventions: Drug: D-Tagatose
- 5.0 mid dose (Active Comparator): 5.0 mid dose - 5.0 g D-tagatose given orally, three times daily, immediately prior to meals for 6 months.
  Interventions: Drug: D-Tagatose
- 7.5 high dose (Active Comparator): 7.5 high dose - 7.5 g D-tagatose given orally, three times daily, immediately prior to meals for 6 months.
  Interventions: Drug: D-Tagatose

INTERVENTIONS:
Drug: D-Tagatose — powder to be dissolved in water prior to dosage.
  Other Names: Naturlose

SUMMARY:
This study is a six-month, prospective, randomized, multicenter, single- blind, controlled clinical study to evaluate the effect of three low-doses of Naturlose (Tagatose) on glycemic control and safety in subjects with Type 2 diabetes under diet control and exercise. The subjects were randomized in one of the 3 arms receiving 2.5, 5 or 7.5 gm of Tagatose.

DETAILED DESCRIPTION:
Screening (Visit 1) and Run-in Period

This period of the study was designed as an 8-week screening and stabilization period, during which potentially eligible subjects participated in a weight-maintaining diet and a daily exercise program.

Subjects who were eligible for screening were diabetic subjects treated solely with diet and exercise and who had mildly elevated HbA1c levels but were otherwise in good health and were not suffering from any serious complications of diabetes.

At the end of the screening visit, potentially eligible study subjects were instructed to follow a weight-maintaining diet and a daily exercise program. They were given a blank subject diary and a nutritional diary, and were scheduled for the second visit (Visit 2) after 8 weeks of stabilization.

Randomization Visit (Visit 2)

At Visit 2, prior to randomization, qualifying study subjects had the following baseline procedures performed: a complete medical evaluation including a review of medical history changes since Visit 1 and a physical examination, blood drawn for clinical laboratory testing.

Randomization was stratified by site and baseline HbA1c levels (< 7.5% or ≥ 7.5%) to obtain a balanced distribution of subjects across the three arms of the trial.

Subjects received a sufficient supply of study medication to last until the next visit. Additionally, the subject received a diary and diary completion instructions for recording side effects, intercurrent illnesses/symptoms, and concomitant medications.

One and Two Month Maintenance Visits (Visit 3 and Visit 4)

At each of these visits, subjects returned to the clinic for diary assessment, blood tests, and study drug compliance assessment and dispensation of additional study drug.

Subjects had blood drawn for clinical laboratory testing including a hematology panel, chemistry panel, creatinine clearance, insulin level, liver function tests, lipid profile, HbA1c level, and urinalysis.

Six Month, End of Study Visit (Visit 5)

During this final visit, all assessments conducted at Visits 3 and 4 were repeated. Additionally, a final physical examination was conducted.

Treatments Administered There were 3 minimal-dose D-tagatose treatment groups in this trial: 2.5 g tid, 5.0 g tid, and 7.5 g tid. The duration of treatment for all groups was 6 months.

Timing of Doses for Each Subject

The tid dosage regimen (i.e., dosing prior to each meal) was selected in order to standardize the fasting status at the time of dose administration across each subjects. The treatment duration of 6 months was determined to be sufficient to evaluate the efficacy and safety of the three dosages for this Phase 2 trial.

DATA QUALITY ASSURANCE

The procedures below were performed to assure the proper conduct of the trial and to assure an accurate, consistent, complete, and reliable report on the data collected during the trial.

Before study initiation and periodically during the study, the monitor visited the investigational sites. A study initiation meeting was held at each investigative site before enrollment of the first subject to review study design, study procedures, data collection, and investigator responsibilities. During interim field monitoring visits, the monitor verified CRF entries against available source documents and ensured that appropriate data were collected and documented. Frequent telephone contact with each study site was maintained throughout the study, and copies of written correspondence between the investigators, sponsor, and IRBs are on file with the sponsor and investigators. Data were collected from the investigational center while respecting the anonymity of all subjects. Prior to data entry, CRFs were checked for completeness and consistency by the monitor and verified against source documentation that was maintained at each study site.

Data from CRF were entered into a relational database (Sequel) via optical character recognition, and subsequently verified versus the CRF by two independent data entry clerks. Any discrepancies in the interpretation of data from the hard copy CRF were referred to a lead data manager who either resolved the discrepancy through review of the CRF or referred the discrepancy to the study site for resolution.

Subsequent to the above data verification processes, programmed validation runs were conducted at regular intervals to check the logic, consistency, and validity of the verified data. Inconsistencies in data logic were referred to the study centers for resolution via data clarification forms (DCF), which required investigator signature.

Data collection and quality assurance/control of electronically transmitted laboratory data were handled according to the respective laboratory's standard procedures before transmission to the CRO for analysis. Programmed validation runs of the central laboratory data versus information from the CRF were performed and discrepancies were reconciled with the study site and the central laboratory.

Prior to data lock for the final analysis, the following quality control procedures were performed.

* An audit of CRF and resolved queries versus analysis data was performed on 100% of the subjects for the primary endpoint, demographics, end of study findings, and randomization information. All errors found during the audit were reported to the lead data manager and corrected.
* An audit of all remaining CRF data (other than primary endpoint, demographics, end of study findings, and randomization information) was performed for a randomly selected 10% of the subjects. If the error rate exceeded 0.5%, a systematic random sampling of an additional 10% of subjects was repeated.

A final audit report and memo summarizing the audit findings was generated and given to the lead data manager and is on file at the CRO.

Data analyses were performed primarily with Statistical Analysis System (SAS®) software, version 9.0 or higher. SAS analysis datasets were crosschecked against the locked database and/or CRF. Data summary tables were crosschecked against SAS analysis datasets. All identified inconsistencies were reported to the lead statistician and resolved prior to production of this report.

This clinical study report was checked for accuracy and consistency before sign-off. This check consisted of a verification of the report text against the report synopsis, and a crosscheck of textual information provided in the report and synopsis versus source summary tables, data listings, and report appendices.

Statistical and Analytical Plan

The CRO prepared a statistical analysis plan (SAP) for the efficacy and safety data before database lock. The SAP was finalized on December 6, 2010.

Analysis Populations

The three analysis populations defined in the SAP, along with their respective definitions and intended use are provided below.

The main efficacy analysis was conducted using the ITT population. The ITT population included all subjects who had signed the ICF, received the protocol-specified treatment, and had a baseline and at least one post-baseline HbA1c value.

The Efficacy Evaluable (EE) population was used for supportive efficacy analyses. The EE population consisted of all randomized subjects who completed the 6-month treatment period, and had no major protocol violations or eligibility violations. All protocol violations were identified prior to breaking the blind.

The safety population consisted of all randomized subjects who received at least one dose of study medication and had at least one post-treatment visit for safety assessment. This population was used for all safety summaries.

Statistical Method Details

Data summaries were prepared for each treatment group and the population as a whole (i.e., all treatment groups combined). The descriptive statistics provided in data summary tables involving continuous data included the number of observations, mean, standard deviation, median, and minimum and maximum values. The descriptive statistics provided in data summary tables involving categorical data included frequency counts and percentages. Inferential statistics were provided only for efficacy endpoints.

Duration of Exposure to Study Drug

The duration (days) of study drug dosing was estimated and summarized descriptively for the Safety Population by dose group and for all doses combined. Duration was based on entries in the CRF and was calculated as last dose date minus first dose date plus one day [(last dose date - first dose date) + 1 day]. If the medication stop date was missing or if the stop date was specified as continuing, the end of study date, as recorded in the CRF, was used as the stop date for duration determination.

Compliance

Percent compliance with study medication was calculated as [(total units of drug returned minus the total units of drug dispensed) ÷ by the total dispensed] times 100%. Resulting data were summarized descriptively for the Safety population by dose group and for all doses combined.

Efficacy Analyses

All efficacy endpoints were summarized descriptively by dose group and for all doses combined for the ITT and the EE populations. All statistical tests for comparisons of dose groups were two-sided tests, with no p-value adjustment. The ITT and EE populations were used in the analyses of efficacy.

Safety Analyses

The Safety Population was used for all analyses of safety and tolerability. All safety parameters were presented descriptively and as data listings. No inferential statistics were planned or performed on safety data.

Adverse Events:

The number and percentage of subjects who reported AE were summarized descriptively by MedDRA System Organ Class (SOC) and Preferred Term (PT), Version 10.0, and dose group. Adverse events and SAEs occurring between randomization and the last study visit are summarized. Unless otherwise specified, the incidences of unique events are provided in all AE summarizations (i.e., a subject is counted only once for each unique event occurring in the summary). For summaries of AEs by severity, if a subject had more than one event per MedDRA SOC or PT, the worst severity was tabulated. Similarly, for summaries of AEs by causality, if a subject had more than one event per MedDRA SOC or PT, the worst severity was tabulated. Additionally, a summary of AEs leading to study drug discontinuation is provided.

Hypoglycemic Episodes:

All subjects experiencing one or more events that coded to the MedDRA PT of "hypoglycemia" were included in the summaries of AEs (see above).

Gastrointestinal Side Effects: Categorical summaries of responses to each of the questions on the GSRS were prepared based on time point and dose group. Additionally, all subjects experiencing one or more events that coded to the MedDRA SOC of "Gastrointestinal Disorders" were included in the summaries of AEs (see above).

Determination of Sample Size

The sample size calculation was based on a reduction of at least 0.5% in HbA1c level after 6 months of the study treatment compared to baseline for each dose group, a standard deviation of 1.0 for each treatment group, and an 80% statistical power with a two-sided analysis at a Type I error rate of 0.05. The required number of evaluable subjects was about 102 (34 for each D-tagatose dose group) based on nQuery Advisor, version 6.01. A total of 40 subjects per treatment group (120 subjects for the study) were to be recruited, as it was expected to observe a 15% drop out rate in this study population, and a total of 150 subjects (50 for per treatment group) was screened based on the estimated screen failure rate of 20%.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics in accordance with WHO.
* Male and female patients, between 18 and 75 years of age.
* Diabetic patients who are not on medication for the disease. Patients may be treated with diet and exercise.
* Normal blood creatine clearance and normal liver function test results.
* BMI less than or equal to 45 kg/m2

Exclusion Criteria:

* Treatment with sulfonylurea (e.g., Glyburide, Glipizide, Glimepiride, Chlorpropamide, Tolazamide, Acetohexamide, or Tolbutamide), TZDs, metformin, acarbose, Byetta, insulin, and any antidiabetic medications within the prior 3 months.
* Therapy with beta-blockers or thiazide diuretics within the prior 3 months
* Pregnancy, breastfeeding, or intention of becoming pregnant or judged to be using inadequate contraceptive measure.
* Documented gastrointestinal disease, or taking of medications likely to alter gut motility or absorption.
* Receiving any investigational drug within 30 days of the baseline visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lodder, Study Director — University of Kentucky
Locations (13):
- United States (5):
  - Probe Clinical Research Corp., Garden Grove, California
  - Pharmax Research Clinic, Miami, Florida
  - PMI Health Research Group, Atlanta, Georgia
  - Ialim Clinical Research Center, Decatur, Georgia
  - Juno Research, LLC, Houston, Texas
- India (8):
  - Diabetes Care and Research Centre, Patna, Bihar
  - Bharti Research Institute of Diabetes and Endocrinology, Karnāl, Haryana
  - Bangalore Endocrinology and Diabetes Research Centre, Bangalore, Karnataka
  - Medisys Clinisearch India Pvt. Ltd., Bangalore, Karnataka
  - Belgaum Diabetes Centre, Belagavi, Karnataka
  - Krishna Diabetes Clinic and Educational Research Centre, Bhopal, Madhya Pradesh
  - Diabetes Thyroid Hormone Research Institute Pvt. Ltd, Indore, Madhya Pradesh
  - Research Health Institute in Diabetes Endocrinology and Metabolism, Mumbai, Maharashtra

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study evaluated the data from 18 clinical study sites (11 sites in the United States and 7 sites in India)for approximately six months.
Pre-assignment Details: Clinical laboratory testing (including comprehensive hematology, clinical chemistry, liver function tests, lipid profile, HbA1c levels and urinalysis) was performed. A urine pregnancy test was performed for female subjects of childbearing potential.
Groups:
- 2.5 Active: Low dose, 2.5 g TID premixed with drinking water into a solution of 4 oz per dose.
- 5.0 Mid Dose: 5.0 dose, 5.0 g TID premixed with drinking water into a solution of 4 oz per dose.
- 7.5 High Dose: high dose. 7.5 g TID premixed with drinking water into a solution of 4 oz per dose.
Period: Overall Study
Arm/Group | 2.5 Active | 5.0 Mid Dose | 7.5 High Dose
Started | 57 | 51 | 53
Completed | 35 | 32 | 34
Not Completed | 22 | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 Active | 5.0 Mid Dose | 7.5 High Dose | Total
Number analyzed (Participants) | 52 | 46 | 47 | 145
Age, Customized [Mean (Standard Deviation); unit: years] — Baseline participants are those from the safety population.
  years
    Age, Continuous | 53.1 (10.2) | 51.1 (11.1) | 51.8 (12.3) | 52.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline participants are from the safety population
  Participants
    Female | 22 | 14 | 19 | 55
    Male | 30 | 32 | 28 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline HbA1c After Six Months of Treatment in Patients With Type 2 Diabetes Mellitus
Description: The primary efficacy parameter was a dichotomous variable: the treatment success as measured by a reduction from baseline HbA1c by at least 0.5 units after six months of treatment (i.e.,0.5% reduction in HbA1c after six months of treatment).
Time Frame: 6 months from baseline
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | 2.5 Active | 5.0 Mid Dose | 7.5 High Dose
Number analyzed (Participants) | 52 | 46 | 47
participants | 10 | 7 | 12
Statistical Analysis 1: Comparison: 2.5 Active vs 5.0 Mid Dose vs 7.5 High Dose; The HbA1c percent change at each study visit was calculated and then categorized as a binary response (i.e., responders and non-responders) for each subject based on the breakpoint to be used in the endpoint. Inferential statistics were prepared to compare the differences across the three treatments a using logistic regression model with the dose group and the HbA1c stratum included in the mode; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = 0.5, Standard Deviation 1.0

2. Secondary Outcome: Effects of Naturlose (Tagatose) on Other Glycemic Control Measurements Such as Plasma Glucose Concentrations and Plasma Lipids at Each Study Visit
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: A Decrease of ≥0.5% in HbA1c Level at Each Study Visit
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: A Decrease of ≥1% in HbA1c Level in Any of the Naturlose (Tagatose) Treatment Groups at Any Time Point Over the Duration of the Study
Time Frame: 8 months
Reporting Status: Not Posted

5. Secondary Outcome: A Decrease of Fasting Plasma Glucose (FPG) Level Compared With Baseline Level at Any Time Point Over the Duration of the Study
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Body Weight Loss (Compared to Baseline)
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: A gastrointestinal Symptom Rating Scale was used. Number of Participants at Risk was based upon the Safety population. Adverse Events were analyzed with regard to the affected organ system only.
Arm/Group | 2.5 Active | 5.0 Mid Dose | 7.5 High Dose
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/46 | 2/47
Other Adverse Events (participants affected / at risk) | 30/52 | 24/46 | 27/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 Active (N=52) | 5.0 Mid Dose (N=46) | 7.5 High Dose (N=47)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia with Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2.5 Active (N=52) | 5.0 Mid Dose (N=46) | 7.5 High Dose (N=47)
Gastrointestinal disorders (Gastrointestinal disorders) | 23 | 16 | 17
Infections and infestations (Infections and infestations) | 10 | 7 | 8
General disorders and administration site conditions (General disorders) | 5 | 5 | 3
Metabolism and Nutrition disorders (Metabolism and nutrition disorders) | 3 | 4 | 5
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4
Nervous system disorder (Nervous system disorders) | 5 | 3 | 3
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No